CLINICAL TRIAL: NCT03516149
Title: The Acute Effect of Foam Rolling on Elbow Joint Sensorimotor Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Fatma Özden, PT, Physical Therapist, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3470-GOA
Record Dates: First submitted 2018-04-24; First posted 2018-05-04 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Proprioceptive Disorders
Keywords: elbow; foam rolling; proprioception; sensorimotor; acute
MeSH Terms: conditions — Somatosensory Disorders

STUDY DESIGN:
Intervention Model Description: There are 2 groups. Study group will receive foam rolling exercise. Control group will receive no foam rolling exercise. They will be handed a brochure about the proprioception and its role in injury prevention and foam rolling . Study group will be evaluated before foam rolling exercise . Afterwards, second evaluation will be performed after exercise at the same day. Control group will be evaluated for the first time. Afterwards, second evaluation will be performed after resting period (2 minutes) at the same day.
Who Masked: Participant
Masking Description: All of participants must be healthy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foam Rolling Group (Experimental): The participants in this group will receive foam rolling exercise.
  Interventions: Other: Foam Rolling Exercise
- Control Group (No Intervention): The participants in this group will receive no foam rolling. They will only be evaluated.

INTERVENTIONS:
Other: Foam Rolling Exercise — Foam rolling exercise will be performed actively. Participants will use a foam roller for exercise. They will position the foam roller on the chair. Afterwards, they will use their body weights to rub the elbow area (biceps brachii muscle) with this foam. There will be 2 sets and each set will be 1 minute. Single set contains 10 repetitions in 1 minute with 30 seconds resting period between sets
  Arms: Foam Rolling Group

SUMMARY:
The purpose of this study is to investigate the acute effects of foam rolling on elbow joint sensorimotor function with healthy participants . Study group will receive foam rolling exercise. Control group will receive no foam rolling exercise. Control group will be given a brochure including information about proprioception and foam rolling.

DETAILED DESCRIPTION:
There is no information in literature about the effects of foam rolling on elbow joint sensorimotor function. The purpose of this study is to investigate acute effects of foam rolling with healthy participants. Study group will receive foam rolling exercise actively by themselves on elbow.

Foam rolling exercise will be applied 10 times each for 1 minute. These exercise will be performed as 2 sets. After each set will be a resting period for 30 seconds. A total of 1 session will be performed. Second evaluation will be performed after exercise at the same day. Control group will receive no foam rolling exercise. They will be handed a brochure about the proprioception and its role in injury prevention and foam rolling. Control group will be evaluated for the first time. Afterwards, second evaluation will be performed after resting period (2 minutes) at the same day.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above healthy participants
* No pain in elbow area within 6 months and at the time of measurement
* To be able to complete all evaluations and applications to be carried out

Exclusion Criteria:

* Having previous foam rolling and self-myofascial relaxation applications on the target area
* Having acne and similar skin problems, open wounds
* Having upper extremity injury, history of fracture or surgery
* Having any systemic musculoskeletal disease
* Having diagnosis of diabetic mellitus or peripheral neuropathy
* Having osteoporosis diagnosis
* Having any cardiovascular disease
* Having vertigo
* Being pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2018-10-20 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Elbow Proprioception | [Time Frame: Baseline, after 1session foam rolling exercise period and then follow up measurement at the same day]
  Change of elbow joint position sense (with digital inclinometer in degree ) and force match ( hand held dynamometer in kg )

SECONDARY OUTCOMES:
Biceps Brachii Strength | [Time Frame: Baseline, after 1session foam rolling exercise period and then follow up measurement at the same day]
  Change of biceps brachii strength ( hand held dynamometer in kg )
Elbow Sensorimotor Performance | [Time Frame: Baseline, after 1session foam rolling exercise period and then follow up measurement at the same day]
  Change of elbow functional motor performance (push up test, modified pull up test, closed kinetic chain upper extremity stability test )

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi Sevi Yeşilyaprak, Phd, Study Director — Dokuz Eylul University
Locations (1):
- Fatma Özden, Izmir, Bornova, Turkey (Türkiye)

REFERENCES:
- [Derived] Yesilyaprak SS, Ozden F. An acute bout of foam rolling of the biceps brachii does not affect upper extremity sensorimotor function: a randomized trial. BMC Musculoskelet Disord. 2025 Nov 13;26(1):1044. doi: 10.1186/s12891-025-09173-y. PMID 41233773